CLINICAL TRIAL: NCT00196755
Title: An Open Label, Randomized, Parallel Design Study to Investigate the Efficacy and Safety of Sevelamer Hydrochloride (Renagel®) Compared With Calcium Acetate in Peritoneal Dialysis Patients
Brief Title: Study of Safety and Efficacy of Renagel® Compared With Calcium Acetate in Patients With Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REN00304
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Peritoneal Dialysis; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer; calcium acetate

ARMS (2):
- Sevelamer Hydrochloride (Renagel®) (Experimental)
  Interventions: Drug: Sevelamer Hydrochloride (Renagel®)
- Calcium acetate (PhosLo® ) (Active Comparator)
  Interventions: Drug: Calcium acetate (PhosLo® )

INTERVENTIONS:
Drug: Sevelamer Hydrochloride (Renagel®) — Sevelamer hydrochloride three times per day with each meal
  Arms: Sevelamer Hydrochloride (Renagel®)
Drug: Calcium acetate (PhosLo® ) — Calcium acetate three times per day with each meal
  Arms: Calcium acetate (PhosLo® )

SUMMARY:
The purpose of this study is to demonstrate that sevelamer hydrochloride is non-inferior to calcium acetate for the treatment of hyperphosphataemia in patients receiving peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign an informed consent form.
* Men or women aged 18 years of age or older.
* A diagnosis of Chronic Kidney Disease (CKD) and receiving peritoneal dialysis (Continuous cyclical peritoneal dialysis (CAPD), Automated peritoneal dialysis (APD) or Continuous cyclical peritoneal dialysis (CCPD) for 8 weeks or longer.
* In the opinion of the investigator, expected to receive peritoneal dialysis for the duration of the study.
* Will have a serum phosphorus level >1.76 mmol/L(5.50 mg/dL) after 2 weeks washout from their usual phosphate binder.
* Will have serum calcium measurement adjusted for albumin within the range (2.10-2.60 mmol/L (8.40-10.40 mg/dL) following 2 weeks washout from their usual phosphate binder.
* Willing to maintain the prescribed sevelamer or calcium acetate for the duration of the study.
* Considered compliant with phosphate binders and dialysis.
* On a stable doses of medication to treat hyperparathyroidism (Vitamin D or its analogues or calcimimetic agents) for the month prior to screening.
* Willing to discontinue use of antacids containing calcium, aluminium or magnesium at screening visit for the duration of the study (unless taken as an evening calcium supplement as prescribed by the investigator per protocol).
* Willing to avoid intentional changes in diet such as fasting or dieting.
* If female and of childbearing potential (pre-menopausal and not surgically sterile), willing to use an effective contraceptive method throughout study, which includes barrier methods, hormones, or Intrauterine devices (IUDs).
* Have a level of understanding and willingness to cooperate with all visits and procedures as described by the study personnel.

Exclusion Criteria:

* Patients with a history of peritonitis in the last 30 days or > 2 episodes in the last 12 months
* Patient with active dysphagia, swallowing disorder, bowel obstruction, or severe gastrointestinal motility disorder.
* Patients who in the opinion of the investigator have poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, Human Immunodeficiency Virus (HIV) infection, or any clinically significant, unstable medical condition.
* Patients with any evidence of active malignancy except for basal cell carcinoma of the skin. A history of malignancy is not exclusion.
* Current use of an antiarrhythmic medication such as quinidine, procainamide, tocainide, or amiodarone for the control of arrhythmias.
* Current use of a seizure medication such as phenytoin, phenobarbital, valproate, or carbamazepine for the control of a seizure disorder.
* Active ethanol or drug abuse, excluding tobacco use.
* If female, are pregnant, planning on becoming pregnant in the next 6 months or breast-feeding.
* Patients with a known hypersensitivity to sevelamer or any constituents of either study drug.
* Patients who have participated in a study of an investigational drug/device during the 30 days preceding the start of the screening period.
* Patients who have any other condition, which in the opinion of the investigator will prohibit the patient's participation in the study.
* Patient is unable to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2004-12; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Compare the effects of sevelamer dosed three times per day (TID) and calcium acetate dosed TID on serum phosphorus. | 12 weeks

SECONDARY OUTCOMES:
Serum calcium- phosphorus (CaxPO4) product | 12 weeks
Serum lipids - total and LDL cholesterol, non- HDL cholesterol, HDL, triglycerides | 12 weeks
Plasma biomarkers: random blood glucose, glycosylated haemoglobin, bone specific alkaline phosphatase, uric acid and c-reactive protein | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (17):
- UZ Gasthuisberg, Leuven, Belgium
- Denmark (3):
  - Aarhus University Hospital, Århus N
  - Fredericia Sygehus, Fredericia
  - Copenhagen University Hospital, Herlev
- CHRU Clémenceau, Caen, France
- Italy (2):
  - Ospedale civico e benfratelli, Palermo
  - Ospedale San Bortolo, Vicenza
- AMC, Amsterdam, Netherlands
- Spain (2):
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
- United Kingdom (7):
  - University Hospital ,Queen Elizabeth Hospital, Birmingham
  - High Wycombe Hospital, Buckinghamshire
  - University of Wales College of Medicine, Cardiff
  - Glasgow Western Infirmary, Glasgow
  - Royal Hospital The Royal London, London
  - Milton Keynes General Hospital, Milton Keynes
  - The Churchill Hospital, Oxford Radcliffe Hospitals NHS Trust, Oxford